CLINICAL TRIAL: NCT01741896
Title: Can Remote Ischaemic Preconditioning Reduce Contrast Induced Nephropathy in Patients Receiving Contrast for Computed Tomography?
Acronym: CT RIPC CIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Stewart Walsh, Professor Stewart Walsh, Mid Western Regional Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Feeley01
Record Dates: First submitted 2012-12-04; First posted 2012-12-05 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Contrast Induced Nephropathy; Remote Ischaemic Preconditioning

ARMS (2):
- RIPC (Active Comparator): Patients in the RIPC arm will undergo a period of upper limb ischaemic preconditioning before their contrast enhanced CT scan. The RIPC stimulus involves four cycles of ischaemia/reperfusion (5 minutes of blood pressure cuff induced upper limb ischaemia with 3 minutes reperfusion). This will start at a time of 30 - 40 minutes before the administration of contrast. The cuff is inflated to 15mmHg above systolic pressure at each inflation.
  Interventions: Procedure: Remote ischaemic preconditioning
- Control arm (No Intervention): Patients in the control arm will undergo no extra intervention.

INTERVENTIONS:
Procedure: Remote ischaemic preconditioning — The intervention is 4 cycles of upper limb ischaemic preconditioning. Each cycle consists of 5 minutes of blood pressure cuff induced ischaemia with 3 minutes of reperfusion. The ischaemic stimulus is induced by inflation of the cuff to 15mmHg above systolic pressure. The reperfusion stimulus is induced by cuff deflation. The RIPC stimulus is commenced at between 30-40 minutes prior to the administration of the IV contrast.
  Arms: RIPC

SUMMARY:
Computated tomography (CT) is an invaluable medical resource for both physicians and surgeons. Contrast media are an aid to improve the diagnostic yield of CT. While an incredibly powerful means of imaging the human body, there are possible complications to the use of contrast including a hypersensitive response and contract induced nephropathy (CIN). The latter will typically occur 48-72 hours after administration.

One recent meta - analysis of serum creatinine levels following contrast enhanced CT found 6.4% of those undergoing this investigation developed CIN. Although typically transient, 1 % had a persisting reduced renal function, with a small minority needing renal replacement therapy (RRT). The development of CIN was influenced by co morbidities and by the amount of contrast given.

The mechanism of injury to the kidney is not definitively established, but is thought most likely due to hypoxia resulting from reduced blood flow, thereby giving rise to oxygen free radicals causing direct damage to the kidney and also direct tubular damage.

Remote conditioning ischaemia has been hypothesized to be nephroprotective, whereby induced transient ischaemia at another site could buffer the impact of the contrast medium's effects. This was first demonstrated during cardiac angiograms, with those patients whom received multiple balloon inflations in the coronary arteries were found to have a lower incidence of CIN than those with fewer balloon inflations. Thus it could be hypothesised that any ischaemia temporarily induced could be nephroprotective. This can be at a point of extremity, rather than involving central organs, such as the arm, with ischaemia induced by the use of a blood pressure cuff, inflated to above systolic blood pressure levels.

No studies have been found in the literature attempting to demonstrate this effect in relation to contrast CT studies. Consequently, a randomised control clinical trial of patients to assess the effectiveness of remote ischaemic preconditioning is proposed.

Study Hypothesis: That performing remote ischaemic preconditioning on those undergoing CTs involving IV contrast is nephroprotective.

ELIGIBILITY:
Inclusion Criteria:

* Hospital inpatients undergoing contrast enhanced abdomino-pelvic CT scanning.

Exclusion Criteria:

* Those with an allergy/hypersensitivity to the contrast solution
* Those with a Cr of above 150μmol/dL on admission, as is a contraindication to IV contrast.
* Patients who are not getting IV contrast
* Any patients with a history of renal transplantation
* Any patients with a history of previous acute kidney injury necessitating management by a nephrologist
* Patients taking either a sulphonlurea or nicorandil.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in eGFR in those undergoing CT with IV contrast | 48 hours
  The study aims to define the effectiveness in the nephroprotective properties of remote ischaemic preconditioning. The outcome measures are the eGFR at 24 and 48 hours post infusion of IV contrast compared to preinfusion levels, in groups randomised into either undergoing RIPC or a control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Mid Western Regional Hospital, Limerick, Limerick, Ireland

REFERENCES:
- [Background] Walsh SR, Tang TY, Sadat U, Gaunt ME. Remote ischemic preconditioning in major vascular surgery. J Vasc Surg. 2009 Jan;49(1):240-3. doi: 10.1016/j.jvs.2008.07.051. Epub 2008 Oct 1. PMID 18829224
- [Background] Whittaker P, Przyklenk K. Remote-conditioning ischemia provides a potential approach to mitigate contrast medium-induced reduction in kidney function: a retrospective observational cohort study. Cardiology. 2011;119(3):145-50. doi: 10.1159/000330930. Epub 2011 Sep 23. PMID 21952203
- [Derived] Healy DA, Feeley I, Keogh CJ, Scanlon TG, Hodnett PA, Stack AG, Clarke Moloney M, Whittaker P, Walsh SR. Remote ischemic conditioning and renal function after contrast-enhanced CT scan: A randomized trial. Clin Invest Med. 2015 May 31;38(3):E110-8. doi: 10.25011/cim.v38i3.22706. PMID 26026638